CLINICAL TRIAL: NCT02649452
Title: Acute Effects of Vibration on Shoulder Flexibility - Experimental Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manisha Parai (Other)
Collaborators: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Sponsor-Investigator, Manisha Parai, Lecturer, Universiti Tunku Abdul Rahman
Organization: Universiti Tunku Abdul Rahman (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U/SERC/84/2015
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Whole body Vibration
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- vibration (Experimental): Flexibility test of Active Chest Flexibility and Shoulder Reach Flexibility tests will be performed before and after the experiment to determine their improvement in the flexibility of the pectoral muscles. After measuring the flexibility, two stretching exercises of one-arm doorway stretch and office chest stretch will be performed. it will be done twice, 30 second each with 10 second rest in between. After exercise, this group had to undergo vibration exercise by using whole body vibration machine.
  Interventions: Other: vibration
- Exercises (Active Comparator): Flexibility test of Active Chest Flexibility and Shoulder Reach Flexibility tests will be performed before and after the experiment to determine their improvement in the flexibility of the pectoral muscles. After measuring the flexibility, two stretching exercises of one-arm doorway stretch and office chest stretch will be performed. it will be done twice, 30 second each with 10 second rest in between
  Interventions: Other: vibration

INTERVENTIONS:
Other: vibration — vibration will be given using whole body vibration machine. The subject will place both palms on top of the vibration platform with their knee supported on the ground. They need to apply as much pressure on the vibration platform by using their body weight. The whole body vibration machine will be set at the frequency of 30 Hz and the amplitude of 5 mm. They need to hold that position for 1 minute for 3 sets with 1 minute rest in between. The researcher will immediately stop this if the subjects feel dizziness and discomfort

SUMMARY:
Whole body vibration (WBV) can help to improve muscle flexibility by stimulating the neuromuscular functions. But there is a dearth in the literature to prove its effectiveness in improving the flexibility of the upper limb muscles. Therefore the purpose of the study is to determine the effects of vibration on improving upper limb flexibility. This experimental research will be conducted by recruiting participants at the age of 19 to 27 with no histories of injuries on the upper limb. They will be randomly assigned into two groups; experimental (with vibration) and control (no vibration) group. The WBV machine will be used to provide vibration to the upper extremities by placing both palms on the vibration platform. The outcome measure of active chest flexibility and shoulder reach flexibility will be performed pre and post vibration.

ELIGIBILITY:
Inclusion Criteria:

* ages of 19 to 28
* no athletic background

Exclusion Criteria:

* shoulder pain and injury within 12 months, recent back pain and neck pain, recent fever and high blood pressure.

Ages: 19 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Active Chest Flexibility test | one minute
Shoulder Reach Flexibility test | one minute

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia